CLINICAL TRIAL: NCT01138384
Title: A Phase I/II Study of Foretinib in Combination With Lapatinib in Patients With Human Epidermal Growth Factor Receptor 2(HER2)Over-Expressing Metastatic Breast Cancer
Brief Title: Study of Foretinib in Combination With Lapatinib in Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I198
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — GSK 1363089; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Foretinib and Lapatinib (Experimental): Patients will receive foretinib as a continuous oral dose, and lapatinib as a continuous oral dose. Lapatinib will commence on Day1, Cycle 1 and foretinib will commence on Day 3, Cycle 1.
  Interventions: Drug: Foretinib; Drug: Lapatinib

INTERVENTIONS:
Drug: Foretinib — Daily oral dosing at assigned dose beginning day 3 of cycle 1
Drug: Lapatinib — Daily oral dosing at assigned dose beginning day 1 cycle 1.

SUMMARY:
This research is being done because it is not yet known what dose of foretinib in combination with lapatinib can be given safely to patients with breast cancer, nor what type and severity of side effects will result from the combination of the two treatments. This research is also being done because it is not clear if the addition of the new drug foretinib to treatment with lapatinib can offer better results and longer survival than treatment with lapatinib alone.

DETAILED DESCRIPTION:
The purpose of this study is to find the dose of foretinib that can safely be given in combination with lapatinib. This is done by starting at doses of both drugs lower than the usual doses of each when given on their own. Patients are given foretinib and lapatinib and are watched very closely to see what side effects they have and to make sure the side effects are not severe. If the side effects are not severe, then more patients are asked to join the study and are given higher does of foretinib and lapatinib. Patients joining the study later on will get higher doses of foretinib and lapatinib than patients who join earlier. This will continue until a dose is found that causes severe but temporary side effects. Doses higher than that will not be given.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of invasive breast cancer, that is human epidermal growth factor receptor 2 (HER2) positive assessed by FISH or IHC 3+ staining (in accordance with ASCO guidelines) on the basis of the local evaluation of HER2 status.
* Formalin fixed paraffin embedded tissue available for translational studies. Patients entered on the expanded RP2D cohort must have an accessible tumour lesion for biopsy.
* Advanced or recurrent/ metastatic disease incurable with standard therapies.
* During the dose escalation phase patients are not required to have measurable disease, but if they do, it will be recorded and followed. Patients at the expanded RP2D must have measurable disease defined by the RECIST 1.1.
* ECOG performance status 0, 1 or 2.
* Age ≥ 18 years of age.
* Any treatment-related major organ toxicities must be recovered to ≤ grade 1.
* Patients may have had prior chemotherapy for adjuvant and/or for metastatic disease. There is no limit to the number of previous chemotherapy regimens allowed provided patients meet other eligibility criteria. A minimum of 21 days since the last dose of chemotherapy must have elapsed prior to registration.
* Patients may have had prior hormone therapy. There is no limit to the number of previous hormone regimens allowed provided patients meet other eligibility criteria. A minimum of 7 days since the last dose of hormone therapy must have elapsed prior to registration.
* Patients may have had prior therapy with trastuzumab or lapatinib. No prior therapy with a c-Met inhibitor or angiogenesis inhibitor. Other targeted agents permissible provided a minimum of 21 days has elapsed since last day of targeted therapy and registration.
* Patients may have had prior radiation therapy provided the patient has recovered from acute toxic effects of the radiation therapy prior to registration and at least 21 days have elapsed from the day of the last fraction of radiation to the date of registration.
* Previous surgery is permitted provided that wound healing has occurred and at least 14 days have elapsed prior to registration if surgery was major.
* Granulocytes (AGC) ≥ 1.5 x 109/L; Platelets ≥ 100 x 109/L
* Serum creatinine ≤ 1.2 x UNL; Total bilirubin ≤ 1.2 x UNL; AST and ALT ≤ 2 x UNL; Potassium within normal range; Magnesium within normal range
* Left ventricular ejection fraction ≥ 50% demonstrated by MUGA scan or echocardiogram within 28 days prior to registration.
* Women must be post menopausal, surgically sterile or use a reliable form of contraception while on study and for 90 days after discontinuing therapy. Women of childbearing potential must have a pregnancy test taken and proven negative within 7 days prior to registration and must not be lactating.
* Patients who require oral anticoagulants (coumadin, warfarin) are eligible
* Patient consent must be obtained according to local Institutional and/or University Human Experimentation Committee requirements.
* Protocol treatment must begin within 2 working days of patient registration.

Exclusion Criteria:

* History of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≥ 5 years.
* Resting BP consistently higher than, systolic > 150 mmHg and/or diastolic > 100 mmHg (in the presence or absence of a stable dose of anti-hypertensive medication) or poorly controlled hypertension, history of labile hypertension or poor compliance with anti-hypertensive medication.
* Appreciable cavitating or actively bleeding lesions.
* Untreated brain or meningeal metastases. (Patients with neurologically stable and treated brain metastases who have discontinued corticosteroids at least two weeks prior to study registration and have no evidence of cavitation or hemorrhage are eligible).
* Serious cardiac illness or condition including, but not limited to:

  * history of documented congestive heart failure (CHF)
  * systolic dysfunction (LVEF < 50% by MUGA or ECHO)
  * high risk uncontrolled arrhythmias (ventricular tachycardia, high-grade AV-block, supraventricular arrhythmias which are not adequately rate-controlled)
  * unstable angina pectoris requiring anti-anginal medication
  * clinically significant valvular heart disease
  * evidence of transmural infarction on ECG
  * New York Heart Association (NYHA) Class III or IV functional status (see Appendix VIII)
  * Patients with QTc > 450 msec are not eligible
* GI tract disease resulting in an inability to absorb oral medication
* Active or uncontrolled infections, or with serious illnesses or medical conditions which would not permit the patient to be managed according to the protocol are not eligible.
* Known hypersensitivity to the study drugs or their components.
* Potent CYP3A4 inhibitors/inducers (e.g. ketoconazole, carbamazepine) must be discontinued at least 7 days prior to Day 1, Cycle 1.
* Patients on treatment with agents with a known risk of Torsades de Pointes (List #1 http://torsades.org) are not eligible.
* Proliferative diabetic retinopathy, retinal arteritis or hemorrhage.
* History of pulmonary embolus or a deep vein thrombosis diagnosed and/or treated within 6 months prior to registration.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-10-27 (Actual); Primary Completion 2014-05-14 (Actual); Study Completion 2015-02-13 (Actual)

PRIMARY OUTCOMES:
Toxicity, maximum administered dose and the recommended phase II dose | every 4 weeks
  Adverse events will be graded using CTCAE V4.0

SECONDARY OUTCOMES:
Pharmacokinetic evaluation of lapatinib | cycle 1 only
  pharmacokinetic evaluation of lapatinib when administered in combination with foretinib
Preliminary evidence of efficacy | every 8 weeks
  All patients with measurable disease will be evaluated for response and progression using RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Chia, Study Chair — British Columbia Cancer Agency
Locations (5):
- Canada (5):
  - BCCA - Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - McGill University - Dept. Oncology, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chia SK, Ellard SL, Mates M, Welch S, Mihalcioiu C, Miller WH Jr, Gelmon K, Lohrisch C, Kumar V, Taylor S, Hagerman L, Goodwin R, Wang T, Sakashita S, Tsao MS, Eisenhauer E, Bradbury P. A phase-I study of lapatinib in combination with foretinib, a c-MET, AXL and vascular endothelial growth factor receptor inhibitor, in human epidermal growth factor receptor 2 (HER-2)-positive metastatic breast cancer. Breast Cancer Res. 2017 May 2;19(1):54. doi: 10.1186/s13058-017-0836-3. PMID 28464908